CLINICAL TRIAL: NCT06597695
Title: A Ketamine-assisted Group Therapy Intervention for Spanish-speaking Adults With Depression
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Juliana Zambrano, MD, MPH (Other)
Responsible Party: Sponsor-Investigator, Juliana Zambrano, MD, MPH, Psychiatrist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024P002122
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label (Experimental): Open label, single arm study
  Interventions: Drug: Ketamine-assisted psychotherapy

INTERVENTIONS:
Drug: Ketamine-assisted psychotherapy — Ketamine-assisted psychotherapy delivered in a group format

SUMMARY:
This is a pilot clinical trial to assess the feasibility, safety, and preliminary efficacy of ketamine-assisted group therapy for Spanish-speaking adults with depression

ELIGIBILITY:
Inclusion Criteria:

1. Self-identifying Latinx, Spanish-speaking 2. Adults 18-64 years 3. Meet DSM-5 criteria for major depressive disorder as evaluated by study clinician 4. Montgomery-Asberg depression scale (MADRS) score of 20 or above at baseline 4. Participants must have an MGB psychiatrist and primary care provider.

Exclusion Criteria:

1. History of primary psychotic disorder, by history
2. History Bipolar I disorder, by history
3. Unstable complex PTSD, as assessed by study clinician
4. History of dissociative identity disorder
5. History of neurocognitive disorder
6. History of severe and/or recent substance use disorder, by history and as assessed by study clinician after clinical evaluation and interview
7. Uncontrolled hypertension, tachycardia, or unstable cardiopulmonary disease, by history a. Blood pressure on initial screen must be <140/90 mmHg.
8. History of aortic dissection
9. History of myocardial infarction
10. History of aneurysm
11. History of hepatic impairment.
12. History of epilepsy
13. History of prior hypersensitivity to ketamine
14. Body Mass Index greater than 35
15. Body Mass Index less than 18.5
16. Are pregnant, breastfeeding, or planning to become pregnant within 12 weeks of treatment completion
17. Enrolled in other clinical trial for the treatment of depression or other behavioral health diagnosis
18. Inability to provide consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate feasibility of a culturally adapted group-based ketamine intervention for Spanish- speaking adults with depression in a community setting | 1 week post-intervention
  (a) Assess the attendance and adherence rates of participants to the group-based ketamine intervention sessions; (b) Evaluate the feasibility of delivering the intervention sessions as planned, including the preparatory, dosing, and integration sessions; (c) Explore the perceptions and experiences of Spanish-speaking participants regarding the intervention.
To assess the safety of a ketamine-assisted group psychotherapy intervention for Spanish-speaking participants with depression in a community setting. | 1 week post-intervention
  (a) assess safety as obtained through vital monitoring; heart-rate variability (HRV) monitoring, EKG, as measured by a Fitbit. (b) evaluate physical and psychological adverse effects at each study visit.

SECONDARY OUTCOMES:
Investigate the preliminary efficacy of the group-based ketamine intervention on psychiatric symptoms, wellbeing, and health behaviors among Spanish-speaking participants with depression. | 1 and 12 weeks post-intervention
  (a) Assess changes in psychiatric symptom scales pre- and post-intervention using validated assessment tools. (b) Measure changes in wellbeing (social wellbeing, personal wellbeing, spiritual health) pre- and post- intervention through self-report scales. Explore shifts in health behaviors pre-and post-intervention, through self-report and accelerometry measures.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Zambrano, MD, Study Director — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Chelsea, Chelsea, Massachusetts, United States